CLINICAL TRIAL: NCT04698889
Title: Study of the Effects of Ingestion of Natural Human, Natural Cow, and Modified-cow Milk, on Glucose, Amino Acids, Insulin, and Incretin Responses in Humans
Brief Title: Effect of Ingestion of Human, Cow, and Modified-cow Milk, on Glucose and Hormone Responses in Humans.
Acronym: PROLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Tessari Paolo, Professor, MD, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Tessari Protocol 1
Record Dates: First submitted 2020-12-14; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Insulin Tolerance; Hormone; Aminoacidaemia
Keywords: cow milk; human milk; incretins; casein; whey proteins

STUDY DESIGN:
Intervention Model Description: Subjects allocated to receive one or more milk types in random order on different occasions, spaced by at least two weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cow milk (Active Comparator): Administration of natural cow whole milk
  Interventions: Dietary Supplement: natural cow
- Human milk (Active Comparator): Administration of natural human milk
  Interventions: Dietary Supplement: natural human
- Modified cow milk - low protein (Active Comparator): Administration of modified cow milk at low protein content
  Interventions: Dietary Supplement: low protein cow milk
- Modified cow milk - high protein (Active Comparator): Administration of modified cow milk at high protein content
  Interventions: Dietary Supplement: high protein cow milk

INTERVENTIONS:
Dietary Supplement: natural cow
  Arms: Cow milk
Dietary Supplement: high protein cow milk
  Arms: Modified cow milk - high protein
Dietary Supplement: natural human
  Arms: Human milk
Dietary Supplement: low protein cow milk
  Arms: Modified cow milk - low protein

SUMMARY:
Human milk, despite a much lower protein content, is as effective as cow milk on insulin stimulation under iso-lactose conditions. The causes for such a similar potency are unknown. This effect could be due to incretin and amino-acid responses, and/or to milk-protein interactions.In this study the investigators will address the above question(s) by testing, in young healthy volunteers, the effects of natural cow and human milk, as well as of the manipulation of the casein and whey protein content in cow milk, on insulin, C-peptide, GLP-1 and GIP secretion, as well as on circulating amino acids.

DETAILED DESCRIPTION:
Objective: To determine plasma glucose, insulin, C-peptide, glucagon-like polypeptide-1 (GLP-1), glucose-inhibitory-polypeptide (GIP) and amino-acid responses, following administration of human and cow milk, either natural or with experimentally-modified casein and whey-protein content(s).

Design. Young healthy volunteers of both sexes will receive iso-lactose loads (0.36 g lactose / kg body weight) of: natural cow milk; natural human milk; and of cow milk with modified casein and whey protein contents. Blood samples will be frequently collected over 4 hours. Plasma glucose, amino acids, insulin and incretin concentrations will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 yrs
* Both sexes
* Healthy
* In post-absorptive state
* Hemoglobin Hb1c values within normal values.
* Previous regular, moderate physical activity
* Stable body weight and regular dietary habits.

Exclusion Criteria:

* Familial or personal history of diabetes.
* Altered fasting glucose and/ or impaired glucose tolerance.
* Any metabolic, hormonal, hepatic, renal, and cardiovascular disease.
* Current drug treatments

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma insulin and c-peptide | 1 year
  microunits and nanomoles
Plasma GIP: glucose-inhibitory polypeptide and GLP-1: glucagon-like-polypeptide-1 | 1 year
  picomol/L and picogram/mL

SECONDARY OUTCOMES:
Plasma Amino acids | 2 years
  micromol/L

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT04698889/SAP_000.pdf
  • Study Protocol (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT04698889/Prot_001.pdf
  • Informed Consent Form (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT04698889/ICF_002.pdf